CLINICAL TRIAL: NCT04055441
Title: A Study of Pattern of Presentation of Pulmonary Tuberculosis Patients Undergoing Treatment at Assiut University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Hussien kilany, resident doctor, Assiut University
Other Study IDs: pulmonary tuberculosis
Record Dates: First submitted 2019-08-06; First posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the investigator's study is to detect the characteristics, pattern and outcome of pulmonary tuberculosis patients treated at Assiut University Hospital by collecting their demographic, clinical, laboratory and radiological data.

DETAILED DESCRIPTION:
Tuberculosis (TB) is a problem of global importance, it is a medical, social and economic disaster of immense magnitude that is occurring over the world

TB remains one of the major health risks associated with morbidity and mortality. Worldwide, about 10 million TB cases have been reported in 2017, and about 1.57 million cases have died The estimated global average risk of infection is 1%, implying approximately 38 million new infections per year among the previously uninfected population .

In Egypt ,researchers have found evidences of tuberculosis in the Egyptian mummies dating from 3000 to 2400 Before Christ and WHO reported that TB is the most important public health problem after hepatitis C , TB disease can affect any organ, but most commonly occurs in the lungs (70%-80%). Pulmonary TB is the most important form of TB infection, because an infection of the lungs is highly contagious due to the mode of droplet transmission .

Patients with TB usually manifest diverse signs and symptoms that vary with age, sex and the associated socio-environmental as well as host factors .

ELIGIBILITY:
Inclusion Criteria:

* All pulmonary tuberculosis adult patients (age ≥ 18 years) who will attend the outpatient clinic of Chest Department at Assiut University Hospital during 2019 - 2020.

Exclusion Criteria:

* Patients less than 18 ys. loss of patient follow-up . extrapulmonary tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — adult patients (age ≥ 18 years) who will attend the outpatient clinic of Chest Department at Assiut University Hospital during 2019 - 2020.
Study Population: - All pulmonary tuberculosis adult patients (age ≥ 18 years) who will attend the outpatient clinic of Chest Department at Assiut University Hospital during 2019 - 2020.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
sputum smear conversion | baseline
  type of positive sample (spontaneous sputum , induced sputum , bronchoalveolar lavage) , technique used for AFB detection (Ziehl - Neelsen (ZN) staining , GeneXpert , conventional TB culture , non-conventional culture )

SECONDARY OUTCOMES:
sputum culture conversion | baseline
  type of positive sample (spontaneous sputum , induced sputum , bronchoalveolar lavage) , technique used for AFB detection (Ziehl - Neelsen (ZN) staining , GeneXpert , conventional TB culture , non-conventional culture )

OTHER OUTCOMES:
time to sputum conversion | baseline
  type of positive sample (spontaneous sputum , induced sputum , bronchoalveolar lavage) , technique used for AFB detection (Ziehl - Neelsen (ZN) staining , GeneXpert , conventional TB culture , non-conventional culture )

CONTACTS AND LOCATIONS:
Overall Officials: amani omar, professor, Principal Investigator — Assiut University

REFERENCES:
- [Background] Rozenshtein A, Hao F, Starc MT, Pearson GD. Radiographic appearance of pulmonary tuberculosis: dogma disproved. AJR Am J Roentgenol. 2015 May;204(5):974-8. doi: 10.2214/AJR.14.13483. PMID 25905930
- [Background] Simon K. [Primary pulmonary tuberculosis in adults]. Munch Med Wochenschr. 1970 May 22;112(21):999-1003. No abstract available. German. PMID 5310017
- [Background] Pirronti T, Cecconi L, Sallustio G, Meduri A, Macis G. Diagnostic imaging of pulmonary tuberculosis. Rays. 1998 Jan-Mar;23(1):93-114. English, Italian. PMID 9673139
- [Background] Huchon G. [Tuberculous infection and pulmonary tuberculosis in adults]. Rev Mal Respir. 1997 Dec;14 Suppl 5:S49-59. French. PMID 9496591
- [Background] Assao Neino MM, Gagara Issoufou MA, Ouedraogo AR, Marcellin KA, Maizoumbou DA, Mamadou S. [The current situation with sputum positive pulmonary tuberculosis in Niamey (Niger)]. Rev Mal Respir. 2019 May;36(5):578-582. doi: 10.1016/j.rmr.2018.07.009. Epub 2019 Apr 19. French. PMID 31010756
- [Background] Cai EZ, Chua SM, Tan M, Tambyah PA. Tuberculosis care: enhancing directly observed therapy in a peri-urban, low socioeconomic status neighbourhood. Singapore Med J. 2019 Jul;60(7):334-336. doi: 10.11622/smedj.2019072. PMID 31378821